CLINICAL TRIAL: NCT06505759
Title: Evaluation of 2%Bromelain Gel With 0.2%Chlorhexidine Gel as Subgingival Local Drug Delivery Following Scaling and Root Planing in Stage II/III and Grade B Periodontitis -Randomized Control Clinical Trail
Brief Title: Evaluation of 2%Bromelain Gel With 0.2%CHX Gel as Subgingival LDD Following SRP in Stage II/III and Grade B Periodontitis -A RCT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-D012-147453
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1-SRP alone (Active Comparator): control group is treated with SRP alone
  Interventions: Procedure: SRP
- GROUP 2-0.2% BROMELAIN gel (Experimental): test group is treated with bromelain gel
  Interventions: Drug: Bromelain gel
- GROUP 3-0.2% CHLORHEXIDINE gel (Active Comparator): test group is treated with chlorhexidine gel
  Interventions: Drug: chlorhexidine gel

INTERVENTIONS:
Drug: Bromelain gel — bromelain gel is prepared from bromelain capsules in laboratory
  Arms: GROUP 2-0.2% BROMELAIN gel
Drug: chlorhexidine gel — chlorhexidine gel is prepared from mouth wash
  Arms: GROUP 3-0.2% CHLORHEXIDINE gel
Procedure: SRP — Scaling and root planing was done with ultra sonic and hand scaling
  Arms: GROUP 1-SRP alone

SUMMARY:
The current study is a prospective randomised study Evaluation of 2%Bromelain Gel With 0.2%Chlorhexidine Gel as Subgingival Local Drug Delivery Following Scaling and Root Planing in Stage II/III and Grade B Periodontitis

DETAILED DESCRIPTION:
36 sites with periodontal pocket depth measuring 4-6mm were selected. The sites selected were divided into

1. Group I (Control)- 12 sites with Probing depth of ≥5mm treated with scaling and root planing alone.
2. Group II -12 sites with Probing depth of ≥5mm treated with scaling and root planing followed by placement of bromelain gel.
3. Group III -12 sites with Probing depth of ≥5mm treated with scaling and root planing followed by placement of chlorhexidine gel.

periodontal pack was placed and patient was recalled at 1week,4th week and 12th week

ELIGIBILITY:
Inclusion Criteria:

* Patient with have chronic periodontitis in the age group between 30-50 years.
* Patients having ≥20 teeth.

  -.Patients with radiographic evidence of bone loss in atleast two teeth.
* Patients who are systematically healthy.
* Patients with localized pockets with probing depth of ≤ 5mm.
* Patients who are cooperative and able to attend the hospital for regular follow-up.

Exclusion Criteria:

* Patients who have received any surgical or nonsurgical therapy during past 6months
* Pregnant or lactating females.
* Use of systemic antibiotics in the past 6 months.
* Patient who are not willing to give a written informed consent

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Probing pocket Depth (PPD) | 3 months
  measured using a UNC-15 probe (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA
Relative attachment level (RAL) | 3 months
  (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA)

SECONDARY OUTCOMES:
Plaque Index | 3 months
  measured on the tooth surface using a probe
Gingival index | 3 month
  measured on the tooth surface using a probe
Modified Sulcus Bleeding Index | 3 months
  measured on the tooth surface using a probe

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. NALLAGATLA VAMSI VENKATA KRISHNA SAI, Bengaluru, Karnataka, India